CLINICAL TRIAL: NCT06998511
Title: Interdisciplinary Collaborative Care Model Combined With Family Empowerment in Patients With Comorbid Hypertension and Diabetes
Brief Title: Interdisciplinary Collaborative Care Model Combined With Family Empowerment in Comorbid Hypertension and Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xiangyang Central Hospital, Affiliated Hospital of Hubei University of Arts and Science (Other Government)
Responsible Party: Principal Investigator, Qiqi Wu, Principal Investigator, Xiangyang Central Hospital, Affiliated Hospital of Hubei University of Arts and Science
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: No. 2025-068
Record Dates: First submitted 2025-05-06; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Hypertension; Diabetes; Blood Pressure Control; Glucose Control; Psychosocial Adaptation
MeSH Terms: conditions — Hypertension; Diabetes Mellitus | interventions — Methods

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- routine nursing intervention (Other): The control group received routine nursing intervention, including basic drug treatment, diet and exercise guidance, psychological counseling, etc.
  Interventions: Other: routine nursing intervention
- interdisciplinary collaborative care and family empowerment (ICCM-FE) intervention (Other): The observation group received interdisciplinary collaborative care and family empowerment (ICCM-FE) intervention based on the COM-B model on the basis of routine care.
  Interventions: Other: interdisciplinary collaborative care and family empowerment (ICCM-FE) intervention

INTERVENTIONS:
Other: interdisciplinary collaborative care and family empowerment (ICCM-FE) intervention — The observation group received interdisciplinary collaborative care and family empowerment (ICCM-FE) intervention based on the COM-B model on the basis of routine care.
  Arms: interdisciplinary collaborative care and family empowerment (ICCM-FE) intervention
Other: routine nursing intervention — The control group received routine nursing intervention, including basic drug treatment, diet and exercise guidance, psychological counseling, etc.
  Arms: routine nursing intervention

SUMMARY:
The Iinterdisciplinary collaborative care model combined with family empowerment (ICCM-FE) intervention based on the COM-B model can effectively improve blood pressure and glucose control in patients with comorbid hypertension and diabetes, enhance their quality of life and psychosocial adaptation, and significantly increase patient satisfaction with nursing care. This intervention has important clinical application value.

DETAILED DESCRIPTION:
To evaluate the efficacy of an interdisciplinary collaborative care model combined with family empowerment (ICCM-FE) based on the COM-B model in managing comorbid hypertension and diabetes, focusing on its impact on blood pressure, glucose control, and psychosocial adaptation. This prospective randomized controlled trial (RCT) enrolled 187 patients with comorbid hypertension and diabetes from January 2023 to March 2024. Patients were randomly assigned to a control group (n = 93) receiving routine care and an observation group (n = 94) receiving ICCM-FE intervention. Follow-up was conducted over 6 months, assessing blood pressure (SBP and DBP), glucose levels (FPG and HbA1c), quality of life (SF-36 scale), psychosocial adaptation (PAIS-SR scale), and nursing satisfaction (NSNS scale) pre- and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients met the diagnostic criteria for hypertension and diabetes as specified in the 《2020 International Society of Hypertension Global Hypertension Practice Guidelines》and the 《2020 American Diabetes Association (ADA) Standards of Medical Care in Diabetes》 ;
* had at least one caregiver, and both the patient and caregiver had basic communication and comprehension abilities to cooperate with the nursing interventions and complete the questionnaires;
* voluntarily participated in the study and signed an informed consent form;
* complete follow-up records.

Exclusion Criteria:

* severe organ dysfunction or mental illness;
* malignancies, severe cardiovascular events (e.g., stroke, myocardial infarction);
* severe hepatic or renal impairment;
* poor adherence or life expectancy less than 1 year.

Ages: 36 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 187 (Actual)
Dates: Start 2023-01-07 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2024-03-16 (Actual)

PRIMARY OUTCOMES:
Blood Pressure Control | Baseline and 6 months.
  Change in systolic blood pressure (SBP) and diastolic blood pressure (DBP) from baseline to 6 months post-intervention.

SECONDARY OUTCOMES:
Quality of Life (SF-36 Scale) | Baseline and 6 months
  Change in SF-36 scores across eight domains (physical function, mental health, role limitations, etc.) from baseline to 6 months post-intervention.
Psychosocial Adaptation (PAIS-SR Scale) | Baseline and 6 months.
  Change in psychosocial adjustment scores (healthcare orientation, occupational/family environment, psychological stress, etc.) from baseline to 6 months post-intervention.
Self-Efficacy (GSES Scale) | Baseline and 6 months.
  Change in General Self-Efficacy Scale (GSES) scores from baseline to 6 months post-intervention.
Nursing Satisfaction (NSNS Scale) | 6 months.
  Patient satisfaction with nursing care measured using the Newcastle Satisfaction with Nursing Services Scale (NSNS) at 6 months post-intervention.

OTHER OUTCOMES:
Adherence to Intervention | Monthly for 6 months.
  Compliance rates with the interdisciplinary collaborative care model (ICCM-FE) assessed via follow-up attendance and task completion logs.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangyang Central Hospital, Affiliated Hospital of Hubei University of Arts and Science, Xiangyang, China